CLINICAL TRIAL: NCT01564199
Title: Effect of Charcoal on Gastrointestinal Absorption of Salmeterol and Fluticasone Propionate.
Brief Title: Phase I Pharmacokinetic Study (SALBLOCK)
Acronym: SALBLOCK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3106006
Record Dates: First submitted 2012-03-21; First posted 2012-03-27 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-03

CONDITIONS: Healthy Volunteer Study
MeSH Terms: interventions — Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A (Experimental): Salmeterol/fluticasone propionate with concomitant charcoal
  Interventions: Drug: salmeterol / fluticasone propionate
- Treatment B (Experimental): Salmeterol/fluticasone propionate without concomitant charcoal
  Interventions: Drug: salmeterol / fluticasone propionate

INTERVENTIONS:
Drug: salmeterol / fluticasone propionate — 100/1000 μg oral capsule

SUMMARY:
The objective of the study is to assess the extent to which the charcoal prevents the absorption of salmeterol and fluticasone via the GI tract. The assessment will be based on comparing the pharmacokinetic parameter area under the concentration-time curve (AUCt).

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females aged 18-60
* Normal weight at least 50 kg

Exclusion Criteria:

* Evidence of a clinically significant cardiovascular, renal, hepatic, haematological, gastrointestinal, pulmonary, metabolic-endocrine, neurological or psychiatric disease.
* Any condition requiring concomitant treatment (including vitamins and herbal products) or likely to need any concomitant treatment during the study.
* Any clinically significant abnormal laboratory value or physical finding that may interfere the interpretation of study result or constitute a health risk for the subject if he/she participates in the study.
* Known hypersensitivity to the active substance(s) or to the excipients of the drug.
* Pregnant or lactating females.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
The pharmacokinetic parameter Area Under Curve (AUC) time frame: predose and 0:15, 0:30, 0:45, 1:00, 1:20, 1:40, 2:00, 4:00, 6:00, 8:00, 10:00, 12:00 and 24:00 hours post-dose. | 24 hours
  The evaluation of primary pharmacokinetic variable AUCt of this study will be based on statistical methods appropriate for crossover study design.

SECONDARY OUTCOMES:
The pharmacokinetic variables Cmax and tmax time frame: predose and 0:15, 0:30, 0:45, 1:00, 1:20, 1:40, 2:00, 4:00, 6:00, 8:00, 10:00, 12:00 and 24:00 hours post-dose. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mika Scheinin, MD, PhD, Principal Investigator — Clinical Research Services Turku Finland
Locations (1):
- CRST (Clinical Research Services Turku), Turku, Finland